CLINICAL TRIAL: NCT04045236
Title: Rectal Cancer AIMS Academy Clinical Research Network Registry
Brief Title: AIMS Academy Clinical Research Network - Non Metastatic Rectal Cancer Operated on With Curative Intent
Acronym: FUCORE
Status: Withdrawn | Type: Observational
Why Stopped: no pts enrolled
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FUCORE TRIAL
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Non Metastatic Rectal Cancer
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non metastatic rectal cancer: Patients receiving the diagnosis of non metastatic rectal cancer and the indication for a curative treatment will be enrolled in the registry. The study population will consist of all the patients enrolled in the participating centres from the start of the rectal cancer registry on.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Data collection

SUMMARY:
The primary purpose of this registry is to prospectively collect data from different Mini-invasive Colo-rectal Units in Northern Italy with a standardization of the pre-operative, intra-operative and post operative setting for patients operated on for non metastatic rectal cancer with curative intent. The secondary aim is to collect in a registry the compliance to oncological treatments and the oncological outcomes for the same patients

DETAILED DESCRIPTION:
Study parameters

Patients with an histological diagnosis of rectal cancer will undergo pre-operative staging as follow:

* Chest-Abdominal TC scan with e.v. contrast.
* Complete colonoscopy
* Pelvic MRI with e.v. contrast with measurements of all the tumours aspects.
* Endorectal US examination
* Serum level of CEA and CA 19,9 and full nutritional status will be analysed
* Complete oncological and pathological medical history examination.
* Data from place of birth and places where patients lived will be collected.
* Sex and race Charlson Comorbidities Index adjusted for age will be calculated for each patient while Robinson Score will be calculated for aged over 70 patients.

Symptoms at presentation (Haemorrhagic framework ,alvo alteration, pain) will be collected. For Locally advance rectal cancer neo adjuvant chemoradiotherapy will be planned. Grey dose received and total dose of chemotherapy administrated together with eventual toxicity and reasons for non completing the therapy will be collected. Patients will be re-staged with pelvic MRI, endorectal US, colonoscopy. Radiological and endoscopic disease response to neo adjuvant treatment criteria will be noted.

Intraoperative analysed parameters will include :

* time of surgery
* blood loss
* type of analgesia
* type of technique, conversion
* level of IMA ligation
* if splenic flexure lowered down
* type of energy device used
* number and type of cartridge used for rectal stapled line
* size of circular stapler used for the anastomosis
* if loop ileostomy performed Isto-pathological examination will performed according to WHO 2010 guidelines, Quirke score and Dworak grade in patients who will undergo neo adjuvant chemo-radiation therapy will be reported. Mismatch repair proteins will be reported when analysed.

Post operative complication will be described according to Clavien Dindo complication scale. Day of discharge and eventual post discharge complication will be evaluated. Application of an ERAS protocol will be added only for at least 80% of ERAS colo-rectal items satisfied. Indication to eventual adjuvant therapy given within a multidisciplinary setting will be noted. Type of therapy, duration of the treatment and a full description of the compliance to the treatment will be described. Oncological follow up will be performed according to National Comprehensive Cancer Network guidelines. Functional follow up will be done yearly with the Low Anterior Resection Syndrome Score.

ELIGIBILITY:
Inclusion Criteria:

* non metastatic rectal cancer with the indication for a curative treatment

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving the diagnosis of non metastatic rectal cancer and the indication for a curative treatment will be enrolled in the registry. The study population will consist of all the patients enrolled in the participating centres from the start of the rectal cancer registry on.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Disease free survival | at 5 years from surgery
  Survival rate
Over all survival | at 5 years from surgery
  Survival rate
Local recurrences | at 5 years from surgery
  Recurrences rate
Distant recurrence | at 5 years from surgery
  Recurrences rate

SECONDARY OUTCOMES:
Quality of life Scale (QOLS) | at 5 years from surgery
  QOLS CRC-specific questionnaire FACT-C score analisys. QOLS CRC Range: 7 maximum 1 minimum. 7 score represents a better value. FACT-C Range maximum 4 minimum 0. 4 score represents better value.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Undecided